CLINICAL TRIAL: NCT05857683
Title: Extension Pin Block vs Pin Orthosis-extension Block Pinning for Bonny Mallet Fractures
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ankara University (Other)
Responsible Party: Principal Investigator, Malik Kısmet, MD, Ankara University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AnkaraUniHand
Record Dates: First submitted 2023-05-04; First posted 2023-05-12 (Actual); Last update posted 2023-05-12 (Actual); Status verified 2023-05

CONDITIONS: Mallet Finger

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- extension pin block (Active Comparator): this is the technique for mallet finger where 2 pins are used, one for the extension block and other intramedullary for the extension posture
  Interventions: Procedure: cextension pin block
- pin orthosis- extension block pin (Active Comparator): this is the technique for mallet finger where only 1 pin is used for extension block and an orthosis is applied for the extension posture
  Interventions: Procedure: pin orthosis- extension block pin

INTERVENTIONS:
Procedure: cextension pin block — this is the technique for mallet finger where 2 pins are used, one for the extension block and other intramedullary for the extension posture
  Arms: extension pin block
Procedure: pin orthosis- extension block pin — this is the technique for mallet finger where only 1 pin is used for extension block and an orthosis is applied for the extension posture
  Arms: pin orthosis- extension block pin

SUMMARY:
This is a single center prospective study comparing the extension pin block vs pin orthosis-extension block pinning for bonny mallet fractures.

DETAILED DESCRIPTION:
Mallet finger is a fracture of the distal phalanx involving the dorsal articular surface. It is important because it concerns the extensor tendon attachment site. The clinical manifestation of mallet finger formation is active extension loss at the DIP joint. If the injury is not treated and becomes chronic, the DIP passive extension is gradually lost and a hyperextension posture occurs in the PIP joint due to the compensatory swan neck deformity. Non-surgical methods have an important place in the treatment of mallet finger injuries. The indications for surgical treatment of mallet finger injuries are a matter of debate. Conditions that are widely accepted as definite surgical indications are open injury, individuals who cannot work with a splint, the ruptured dorsal part is large and includes more than 30% of the articular surface, and the presence of palmar subluxation in the DIP. Among the mallet finger surgical treatments, the extension pin block technique , bracing in extension, hook method are defined.

In this prospective study, we aimed to compare the extension pin block technique with the pin orthosis-extension block pinning. In comparison, the patients eligible for the study will be evaluated according to Crawford criteria for function evaluation, complications (infection, nail deformities, skin necrosis, DIP joint osteoarthritis), recovery time.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and older patients
* Wehbe classification type 2 b (Type Definition) I No DIP joint subluxation II DIP joint subluxation III Epiphyseal and physeal injuries Subtype A Avulsed fragment <1/3 of articular surface B Avulsed fragment 1/3-2/3 of articular surface C Avulsed fragment >2/3 of articular surface )
* Isolated bonny mallet fractures
* Minimum 1 year follow up
* Good cognitive status

Exclusion Criteria:

* Patients under the age of 18
* Open fracture
* Chronic mallet finger
* TFracture area that includes more than 50% of the joint face
* Patients whose follow-up less than 1 year

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2023-05-01 (Actual); Primary Completion 2024-05-01 (Estimated); Study Completion 2024-06-01 (Estimated)

PRIMARY OUTCOMES:
Crawford criteria | postoperative 1st day
  functional scoring for the DIP joint, focuses on range of motion and pain
Crawford criteria | postoperative 1st month
  functional scoring for the DIP joint, focuses on range of motion and pain
Crawford criteria | postoperative 3rd month
  functional scoring for the DIP joint, focuses on range of motion and pain
Crawford criteria | postoperative 6th month
  functional scoring for the DIP joint, focuses on range of motion and pain
Crawford criteria | postoperative 12th month
  functional scoring for the DIP joint, focuses on range of motion and pain

SECONDARY OUTCOMES:
complications | postoperative 1st day
  skin necrosis, loss of range of motion, infection, nail bed injury
complications | postoperative 1st month
  skin necrosis, loss of range of motion, infection, nail bed injury
complications | postoperative 3rd month
  skin necrosis, loss of range of motion, infection, nail bed injury
complications | postoperative 6th month
  skin necrosis, loss of range of motion, infection, nail bed injury
complications | postoperative 12th month
  skin necrosis, loss of range of motion, infection, nail bed injury

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara University Medical Faculty, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Collected data will be shared after reaching the minimum required number and performing the analysis
Supporting Information: Study Protocol, SAP
Time Frame: June 2024